CLINICAL TRIAL: NCT04444089
Title: Role of Lung Ultrasound in Comparison of Different Fluid Replacement Regimens in Pediatric Patients Undergoing Penile Hypospadias Repair, Randomized Control Trial
Brief Title: Perioperative Fluid Therapy in Pediatric Patients Undergoing Penile Hypospadias Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: N-1 / 2020
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Volume Overload
Keywords: Conventional regimen; restrictive regimen; lactated Ringer's solution; lung ultrasound; fluid management
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional group, CG (Experimental): receives Ringer's lactate solution at a rate of 4 ml/kg/h for the first-10 kg of body weight, 2 ml/kg/h for the second-10 kg of body weight, and 1 ml/kg/h for each further kg of body weight. The deficit volume is calculated as the maintenance volume multiplied by fasting hours and given as follows: 50% of the volume in the first hour, 25% of the volume in the second hour, and 25% of the volume in the third hour, in addition to the aforementioned maintenance volume
  Interventions: Diagnostic Test: lung ultrasound
- restricted group, RG (Experimental): Patients in the RG receives Ringer's lactate solution at a rate of 3 ml/kg/h from the start to the end of surgery.
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — Lung ultrasound with a curvilinear probe (DDED) is performed in all patients in a supine position on the lateral wall of the chest at approximately the level of the lower ribs using an ultrasound probe at a frequency of 4-12 MHz (AcusonX300, Siemens Korea, Seoul, South Korea). The mean number of B-lines detected on the ultrasound image and the percentage of patients who showed B-lines on their images were recorded. The mean of three measurements is used. Inter-observer variability is estimated to be 0.766 (95% confidence interval 0.675-0.847).

SUMMARY:
Optimization of perioperative fluid management is important for preventing adverse events, such as hypovolemia, cardiogenic shock, volume overload, and pulmonary edema, in both adult and pediatric patients. If the intravascular (IV) fluid volume is not optimized, pediatric patients are at risk of dehydration or volume overload. Perioperative IV fluid therapy is important during and after induction of general anesthesia (GA).The aim of this study is to investigate the difference between conventional and restrictive fluid replacement regimens using lung ultrasound in pediatric patients undergoing penile hypospadias repair, as a surgery with minor fluid loss.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for repair of penile hypospadias with American Society of Anaesthesiologists' physical status of class I-II.

Exclusion Criteria:

* Patients with pulmonary, cardiovascular, or hematological disorders or a family history of allergy to local anesthetics or lung disease

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
volume overload using lung ultrasound | intraoperative duration that is approximately 110 minutes.
  volume overload using lung ultrasound according to The mean number of B-lines detected on the ultrasound image

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsonbaty, M.D., Principal Investigator — Cairo University
Locations (1):
- anesthesia department at Cairo University, Cairo, Elmanial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to be shared

REFERENCES:
- [Background] 1. Joshua IS. Perioperative fluid restriction. Clin Colon Rectal Surg 2013;26:197-202. 2. Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, et al. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: Consensus statement for anaesthesia practice. Acta Anaesthesiol Scand 2016;60:289-334. 3. Varadhan KK, Lobo DN. A meta-analysis of randomised controlled trials of intravenous fluid therapy in major elective open abdominal surgery: Getting the balance right. Proc Nutr Soc 2010;69:488-9. 4. Shin CH, Long DR, McLean D, Grabitz SD, Ladha K, Timm FP, et al. Effects of intraoperative fluid management on postoperative outcomes: A hospital registry study. Ann Surg 2018;267:1084-92.